CLINICAL TRIAL: NCT01786733
Title: Psychotherapy in the Transition From Acute Psychiatric Inpatient Wards to Outpatient Services - A Randomized Controlled Trial of Behavioral Activation vs. Supportive Therapy
Brief Title: Behavioral Activation - From Inpatient to Outpatient Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Fredrik Folke, PhD-student, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2012 / 226
Record Dates: First submitted 2013-01-29; First posted 2013-02-08 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Inpatient Facility Diagnoses; Psychiatric Disorders; Depressive Symptoms
Keywords: Acute Inpatient Psychiatry; Continuity of Care; Behavioral Activation; Depression
MeSH Terms: conditions — Mental Disorders; Depression | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Activation (Experimental): Behavioral Activation + Treatment as Usual. 12 sessions twice weekly (i.e. 6 weeks). Individual therapy. Therapy is initiated during inpatient admission and continue after discharge. Protocol aimed at increased activation towards goals and personal values and decreased avoidance behaviors.
  Interventions: Behavioral: Behavioral Activation
- Supportive Therapy (Active Comparator): Supportive Therapy + Treatment as Usual. 12 sessions twice weekly (i.e. 6 weeks). Individual therapy. Therapy is initiated during inpatient admission and continue after discharge. Protocol aimed at providing psychological non-directive support.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation
  Arms: Behavioral Activation
Behavioral: Supportive Therapy
  Arms: Supportive Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of Behavioral Activation and Supportive Therapy added to the standard acute psychiatric inpatient care. Therapy starts during inpatient care and can continue in an outpatient facility if the patients are discharged before 12 sessions has been completed.

DETAILED DESCRIPTION:
Psychiatric inpatient care is reserved for individuals with the most acute mental health problems. The period after discharge is associated with increased risk for relapse, non-adherence and suicide. Delivering high quality psychosocial interventions during and after acute psychiatric inpatient care is known to be a difficult challenge. This study will investigate the effectiveness of adding either Behavioral Activation or Supportive Therapy to the standard acute psychiatric inpatient care. Subjects with different psychiatric diagnoses and elevated depressive symptoms are assessed and randomized after admission. Therapists from the nearest outpatient facility initiate 12 sessions of Behavioral Activation or Supportive Therapy as soon as possible. The 12 sessions are delivered twice weekly at the inpatient unit or at the outpatient facility, depending on whether the patient is admitted or discharged. Treatment as usual interventions(medications, nursing etc.) are not manipulated in the study. The main assessment points are pre-, post, 6 months follow-up and 12 months follow-up. The main outcome measure and some process measures are also administered at session 3, 6 and 9.

ELIGIBILITY:
Inclusion Criteria:

* Admitted into one of four acute psychiatric inpatient units in Dalarna
* MADRS-S 20 and above at acute admission and and after 2-3 days on the ward
* Psychiatric disorder according to M.I.N.I (Sheehan et al., 1998)
* Read and Speak Swedish

Exclusion Criteria:

* Acute psychotic symptoms
* Acute manic symptoms
* Confusion
* Primary eating disorder
* Primary alcohol or substance abuse disorder
* Self rated score on AUDIT (Saunders et al., 1993)of 20 or greater
* Mental retardation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (Self-report version) (MADRS-S) | Weekly during treatment period of 6 weeks
  MADRS-S is a 9 item self report measure of depressive symptoms.
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (Self-report version) (MADRS-S) | 24 hours
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (Self-report version) (MADRS-S) | 6 months
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (Self-report version) (MADRS-S) | 12 months

SECONDARY OUTCOMES:
Change from baseline in EuroQol 5 Dimension Scale (EQ5D) | 24 hours
  The EQ5D is a self rating measure for health-related quality of life. It consists of 5 health state dimensions (mobility, self-care, usual activity, pain/discomfort and anxiety/depression) on which the respondent has to indicate his own health state.
Change from baseline in EuroQol 5 Dimension Scale (EQ5D) | 6 months
Change from baseline in EuroQol 5 Dimension Scale (EQ5D) | 12 months
Change from baseline in Alcohol Disorders Identification Test (AUDIT) | 24 hours
  10 item screening instrument for alcohol use
Change from baseline in Alcohol Disorders Identification Test (AUDIT) | 6 months
  10 item screening instrument for alcohol use
Change from baseline in Alcohol Disorders Identification Test (AUDIT) | 12 months
  10 item screening instrument for alcohol use
Change from baseline in The Sheehan Disability Scale (SDS) | 24 hours
  The SDS is a three-item, self-report scale used to assess functioning in three areas of life (work, social life, and family life). Each item is rated on an 11-point Likert-type scale ranging from zero (no impairment) to 10 (extreme impairment), while the total range extends from zero to 30 points.
Change from baseline in The Sheehan Disability Scale (SDS) | 6 months
Change from baseline in The Sheehan Disability Scale (SDS) | 12 months
Change from baseline in Behavioral Activation for Depression Scale, Short Form (BADS-SF) | 24 hours
  9 item self rating instrument of activation and avoidance.
Change from baseline in Behavioral Activation for Depression Scale, Short Form (BADS-SF) | Weekly druing treatment period of 6 weeks
  9 item self rating instrument of activation and avoidance.
Change from baseline in Behavioral Activation for Depression Scale, Short Form (BADS-SF) | 6 months
  9 item self rating instrument of activation and avoidance.
Change from baseline in Behavioral Activation for Depression Scale, Short Form (BADS-SF) | 12 months
  9 item self rating instrument of activation and avoidance.
Change from baseline in sick leave and employment status | 6 months
  Interview questions regarding Days on/type of/level of sick leave Interview questions regarding employment status and hours of work per week
Change from baseline in sick leave and employment status | 12 months
Change from baseline in Mini-International Neuropsychiatric Interview (M.I.N.I) | 24 hours
  The Mini International Neuropsychiatric Interview is a short, structured interview designed for clinicians to diagnose psychiatric disorders in accordance with the Diagnostic and Statistical Manual (DSM-IV) and International Classification of Diseases (ICD-10).
Change from baseline in Mini-International Neuropsychiatric Interview (M.I.N.I) | 6 months
  The Mini International Neuropsychiatric Interview is a short, structured interview designed for clinicians to diagnose axel I DSM-IV and ICD-10 disorders.
Change from baseline in Mini-International Neuropsychiatric Interview (M.I.N.I) | 12 months
  The Mini International Neuropsychiatric Interview is a short, structured interview designed for clinicians to diagnose axel I DSM-IV and ICD-10 disorders.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours
  Interview for clinician rating of depressive symptoms. 10 items each ranging from 0-6.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 months
  Interview for clinician rating of depressive symptoms. 10 items each ranging from 0-6.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 12 months
  Interview for clinician rating of depressive symptoms. 10 items each ranging from 0-6.
Change from baseline in Global Assessment of Functioning (GAF) | 24 hours
  Clinicians and patients rate severity of symptoms and functioning on a scale ranging from 1-100.
Change from baseline in Global Assessment of Functioning (GAF) | 6 months
  Clinicians and patients rate severity of symptoms and functioning on a scale ranging from 1-100.
Change from baseline in Global Assessment of Functioning (GAF) | 12 months
  Clinicians and patients rate severity of symptoms and functioning on a scale ranging from 1-100.
Change from baseline in Clinical Global Impression (CGI) | 24 hours
  Clinician rates patients' psychiatric problems in regards to severity on a scale from 0-6. After treatment the clinician rates the degree of change in relation to the first assessment.
Change from baseline in Clinical Global Impression (CGI) | 6 months
Change from baseline in Clinical Global Impression (CGI) | 12 months
Change from baseline in Usage of mental health care | 6 months
  Re-admissions (frequency/length of admissions), outpatient visits, usage of psychiatric medications. Data from medical charts.
Change from baseline in Usage of mental health care | 12 months
  Re-admissions (frequency/length of admissions), outpatient visits, usage of psychiatric medications. Data from medical charts.

CONTACTS AND LOCATIONS:
Overall Officials: Per Söderberg, PhD, Study Director — The Adult Psychiatric Clinic of Landstinget Dalarna, Sweden; Lisa Ekselius, Professor, Study Chair — Department of Neuroscience, Psychiatry, Uppsala University, Sweden; Stefan Tungström, PhD, Study Chair — The Adult Psychiatric Clinic of Landstinget Dalarna, Sweden; Timo Hursti, PhD, Study Chair — The Department of Psychology, Uppsala University, Sweden; Fredrik Folke, PhD-student, Principal Investigator — Department of Neuroscience, Psychiatry, Uppsala University, Sweden